CLINICAL TRIAL: NCT01622413
Title: Transforaminal Endoscopic Surgery Cost Outcome Research Trial
Brief Title: Trial to Show Non-inferiority / Superiority of an Endoscopic Transforaminal Discectomy to Standard Microdiscectomy
Acronym: TESCORT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Patients did not consent to randomization in any study center, since they preferred endoscopic surgery. The recruitment of patients was impossible.
Sponsor: Joimax GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/001
Record Dates: First submitted 2012-06-12; First posted 2012-06-19 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Lumbar Disc Herniation
Keywords: lumbar spine; herniated disc; slipped disc; disc herniation; discectomy; nucleotomy; disc surgery; endoscopy; spine
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — TES

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endscopy (Experimental)
  Interventions: Procedure: joimax TESSYS
- Microsurgery (Active Comparator)
  Interventions: Procedure: Microdiscectomy

INTERVENTIONS:
Procedure: joimax TESSYS — Transforaminal Endoscopic Surgery System
  Other Names: TES; TESS
  Arms: Endscopy
Procedure: Microdiscectomy — Standard procedure for disc surgery
  Arms: Microsurgery

SUMMARY:
This study compares an endoscopic transforaminal surgical technique for the treatment of a herniated disc to the standard microsurgical procedure. Clinical parameters as well as health economy will be assessed.

The study hypothesis is that the endoscopic approach is equivalent or superior to microdiscectomy.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic lumbar disc herniation
* clinical and radiological evidence of nerve root compression
* failure of conservative treatment for at least 6 weeks

Exclusion Criteria:

* previous lumbar spine surgery
* severe or progressive motor deficit
* BMI > 40
* cauda equina syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2017-01 (Estimated); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Oswestry Disability Index at 4 years | total follow-up period of 4 years

SECONDARY OUTCOMES:
Change from baseline in Quality of Life (SF-12) | total follow-up period of 4 years
Health resources consumption | total follow-up period of 4 years
Complication rate | 2 years
Patient satisfaction | Total follow-up period of 4 years
Change from baseline in back and leg pain (NRS) | total follow-up period of 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Carl H Fürstenberg, MD, Principal Investigator — University Clinic Heidelberg, Department of Orthopedics, Traumatology and Paraplegiology
Locations (3):
- University Clinic of Neurosurgery, Graz, Austria
- Germany (2):
  - Ligamenta Spine Center, Frankfurt
  - University Clinic Heidelberg, Department of Orthopedics, Traumatology and Paraplegiology, Heidelberg